CLINICAL TRIAL: NCT06157437
Title: An Exploratory Study of Focal Pulse Ablation System in the Treatment of Atrial Arrhythmia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Dinova EP Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fPFA001
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Typical Atrial Flutter; Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Focal pulse ablation system (Experimental)
  Interventions: Device: Focal Pulse field Ablation

INTERVENTIONS:
Device: Focal Pulse field Ablation — Bidirectional block of the cavo-tricuspid isthmus (CTI) was performed with the novel focal pulse field ablation.

SUMMARY:
This is a prospective, single-group clinical study. The objective is to evaluate the safety and efficacy of focal pulse ablation system in the treatment of typical atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged at least 18;
* Subjects with at least one typical atrial flutter attack recorded by ECG or holter in the 180 days prior to enrollment, and the ECG of other hospitals could be accepted;
* Subjects are able to understand the purpose of the study, voluntarily participate in the study and sign the informed consent, and are willing to complete the follow-up according to the requirements of the program.

Exclusion Criteria:

* Any prior cavo-tricuspid isthmus ablation;
* Unstable angina;
* Atrial flutter secondary to electrolyte disorder, thyroid disease or other reversible causes;
* Myocardial infarction or coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) within the prior three months;
* At baseline, New York College of Cardiology (NYHA) heart function grades III and IV;
* Implantable devices such as ICDs, CRTS and pacemakers in the body;
* Atrial or ventricular tumors, blood clots, thrombus, or known clotting disorders were recorded within the prior 90 days;
* Severe structural heart disease, including tricuspid stenosis, tricuspid malformation, or other congenital heart disease that prevents ablation surgery;
* Previously received tricuspid metal valve replacement;
* Thromboembolic events (including transient ischemic attacks) within the past 6 months;
* Mural thrombosis, tumor, or other abnormality that interferes with vascular puncture or catheter operation;
* Severe lung disease, pulmonary hypertension or any lung disease involving abnormal blood gas or severe breathing difficulties;
* Anticoagulation contraindications and a history of blood clotting or abnormal bleeding;
* Acute systemic infection;
* Serum creatinine greater than twice the upper limit of normal, or any history of renal dialysis;
* Women who are pregnant or breastfeeding or who cannot use contraception during the study period;
* Enrollment in another clinical trial evaluating other devices or drugs during the same period;
* Life expectancy less than 12 months (e.g. advanced malignancy);
* Abnormalities or diseases considered by the investigator to be excluded from inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute procedural success | immediately after the procedure
  Acute procedural success is defined as the creation of bidirectional conduction block across the cavo-tricuspid isthmus immediately and 30 minutes after ablation.

SECONDARY OUTCOMES:
Chronic success | 6 months after procedure
  Chronic success is defined as the absence of recurrent atrial flutter at 6 months post-ablation according to electrocardiogram data, including electrocardiogram, 24-hour Holter.
Ablation efficiency including total procedure time, catheter dwell time, pulse discharge time and total X-ray exposure time | immediately after the procedure
  Total procedure time (defined as the total time from initial femoral venipuncture to final catheter removal), catheter dwell time (time between the pulsed field ablation catheter entering the left atrium and its withdrawal from the left atrium), pulse discharge time (The total time of delivering pulse energy through the pulsed field ablation catheter, single ablation time ablation times), total X-ray exposure time (the total time of X-ray imaging of the catheter)
Incidence of device-related major adverse events (MAE) within 7 days after ablation | within 7 days after ablation
  Device-related MAE includes death, myocardial infarction, pulmonary embolism, stroke /TIA, severe pericardial effusion, and complete atrioventricular block.
Incidence of device-related severe adverse events (SAE) | 3 months and 6 months after procedure
  Device-related SAE refers to a device-related event that occurs during the clinical trial that results in mortality or serious deterioration in patient health, including a fatal illness or injury, a permanent defect in body structure or body function, or an event that requires medical or surgical intervention to avoid one or more permanent defects in body structure or body function.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No